CLINICAL TRIAL: NCT01361308
Title: A Phase 3, Twelve-Week, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Efficacy and Safety Study of Mesafem (Paroxetine Mesylate) Capsules in the Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: Efficacy/Safety Study of Brisdelle™ (Formerly Known as Mesafem) in the Treatment of Vasomotor Symptoms (VMS)
Acronym: N30-003
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N30-003
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Postmenopausal Symptoms
Keywords: Menopause; Vasomotor Symptoms; Hot Flashes Perimenopause; Climacteric Symptoms; Mesafem; Low-Dose Mesylate salt of Paroxetine (LDMP)
MeSH Terms: interventions — Paroxetine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brisdelle (paroxetine mesylate) (Experimental): Brisdelle (paroxetine mesylate)
  Interventions: Drug: Brisdelle (paroxetine mesylate)
- Placebo Capsules (Placebo Comparator): Placebo Capsules
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Brisdelle (paroxetine mesylate) — Subjects will be randomized to receive either Brisdelle (paroxetine mesylate) Capsules 7.5 mg or placebo in a 1:1 ratio, administered once daily at bedtime beginning on Day 1 and continuing up to Day 84
  Other Names: Former Names: Mesafem Capsules or; LDMP (Low-Dose Mesylate salt of Paroxetine)
  Arms: Brisdelle (paroxetine mesylate)
Drug: Placebo capsules — Subjects will be randomized to receive either Brisdelle (paroxetine mesylate) Capsules 7.5 mg or placebo in a 1:1 ratio, administered once daily at bedtime beginning on Day 1 and continuing up to Day 84
  Other Names: Sugar pill
  Arms: Placebo Capsules

SUMMARY:
The purpose of this study is to assess the safety & efficacy of Brisdelle (paroxetine mesylate) Capsules 7.5 mg for treatment of vasomotor symptoms (VMS) associated with menopause.

DETAILED DESCRIPTION:
This is 12-week, multicenter, double-blind, randomized, placebo-controlled study of Brisdelle (paroxetine mesylate) Capsules 7.5 mg and placebo capsules in subjects with moderate to severe postmenopausal VMS, defined as follows:

* Moderate VMS: Sensation of heat with sweating, able to continue activity
* Severe VMS: Sensation of heat with sweating, causing cessation of activity

The study is comprised of a screening period, a run-in period, a baseline visit, and a double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Female, ≥ 40 years of age at screening (inclusive)
2. Reported more than 7-8 moderate to severe hot flashes per day (average) or 50-60 moderate to severe hot flashes per week for at least 30 days prior to the screening visit
3. Spontaneous amenorrhea for at least 12 consecutive months or
4. Amenorrhea for at least 6 months and meet the biochemical criteria for menopause or
5. Bilateral salpingo-oophorectomy ≥ 6 weeks with or without hysterectomy

Exclusion Criteria:

1. Known non-responder to previous Selective serotonin reuptake inhibitor (SSRI) or Serotonin norepinephrine reuptake inhibitor (SNRI) treatment for VMS
2. History of self injurious behavior
3. History of clinical diagnosis of depression or treatment for depression
4. History of clinical diagnosis of borderline personality disorder
5. Use of an investigational study medication within 30 days prior to screening or during the study
6. Concurrent participation in another clinical trial or previous participation in this trial
7. Family of investigational-site staff

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Jacobs, MD, Principal Investigator; Donna DeSantis, MD, Principal Investigator; Robert Phillips, MD, Principal Investigator; Louise Taber, MD, Principal Investigator; Paige C. Brainard, MD, Principal Investigator; Mark Stripling, MD, Principal Investigator; Gioi Smith-Nguyen, MD, Principal Investigator; Anthony Dulgeroff, MD, Principal Investigator; Elise Kwon, MD, Principal Investigator; Douglas Young, MD, Principal Investigator; William Koltun, MD, Principal Investigator; Dana Shipp, MD, Principal Investigator; Eric Ross, MD, Principal Investigator; Arthur Waldbaum, MD, Principal Investigator; Theodore Cooper, MD, Principal Investigator; J B. Stern, MD, Principal Investigator; Paul DiGrazia, MD, Principal Investigator; Robert Spitz, MD, Principal Investigator; James A Simon, MD, Principal Investigator; Mildred Farmer, MD, Principal Investigator; James Andersen, MD, Principal Investigator; Steven Bowman, MD, Principal Investigator; Rene Casanova, MD, Principal Investigator; Mary Yankaskas, MD, Principal Investigator; Andrew Kaunitz, MD, Principal Investigator; Ronald Surowitz, MD, Principal Investigator; Lisa Cohen, MD, Principal Investigator; Lisa Vendeland, MD, Principal Investigator; Tyrone Malloy, MD, Principal Investigator; Stephen C. Blank, MD, Principal Investigator; Mark Turner, MD, Principal Investigator; Carl R Lang, MD, Principal Investigator; Arthur Donovan, MD, Principal Investigator; Armen Arslanian, MD, Principal Investigator; Shiao-Yu Lee, MD, Principal Investigator; Gayle Moyer, MD, Principal Investigator; Geoffrey Turner, MD, Principal Investigator; Susan L Hendrix, MD, Principal Investigator; Mark Barber, MD, Principal Investigator; Stephen Swanson, MD, Principal Investigator; Timothy Sauter, MD, Principal Investigator; Steven Sussman, MD, Principal Investigator; Elizabeth Bretton, MD, Principal Investigator; Lance A. Rudolph, MD, Principal Investigator; Kenneth Levey, MD, Principal Investigator; Pouru Bhiwandi, MD, Principal Investigator; Richard E. Hedrick, MD, Principal Investigator; Gregory P Tarleton, MD, Principal Investigator; Mira Baron, MD, Principal Investigator; David J Portman, MD, Principal Investigator; Milroy Samuel, MD, Principal Investigator; Stuart Weprin, MD, Principal Investigator; James Liu, MD, Principal Investigator; Angelique Barreto, MD, Principal Investigator; Marvin Kalafer, MD, Principal Investigator; Larry S. Seidman, MD, Principal Investigator; Saul R. Berg, MD, Principal Investigator; Susan Floyd, MD, Principal Investigator; Scott Wilson, MD, Principal Investigator; Cynthia Strout, MD, Principal Investigator; D. S. Harnsberger, MD, Principal Investigator; Janet Dittus, MD, Principal Investigator; Gregg Lucksinger, MD, Principal Investigator; Anna Damian, MD, Principal Investigator; Sandra Hurtado, MD, Principal Investigator; Alfred Poindexter, MD, Principal Investigator; Nancy Campbell, MD, Principal Investigator; William Jennings, MD, Principal Investigator; Jose Ruiz, MD, Principal Investigator; John A. Hoekstra, MD, Principal Investigator; Peter A. Zedler, MD, Principal Investigator; Franklin Morgan, MD, Principal Investigator; Robin Kroll, MD, Principal Investigator; Derrick R Havin, MD, Principal Investigator
Locations (74):
- United States (74):
  - Wilmax Clinical Research, Mobile, Alabama
  - East Valley Family Physicians PLC, Chandler, Arizona
  - Advanced Research Associates, Glendale, Arizona
  - Premier Research Group Limited, Peoria, Arizona
  - Verona Clinical Research, Inc, Tucson, Arizona
  - NEA Baptist Women's Clinic, Jonesboro, Arkansas
  - Grossmont Center for Clinical Research, La Mesa, California
  - High Desert Medical Group, Lancaster, California
  - Facey Medical Foundation, Mission Hills, California
  - Northern California Research, Sacramento, California
  - University Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Apex Research Institute, Santa Ana, California
  - Downtown Women's Health Care, Denver, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - The Women's Clinic of Northern Colorado, Fort Collins, Colorado
  - Danbury Clinical Research, LLC, Danbury, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - James A. Simon, MD, PC, Washington D.C., District of Columbia
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - DBC Research, Deerfield Beach, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - University of Florida College of Medicine - Jacksonville Southside Women's Health, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Affinity Healthcare, Arlington Heights, Illinois
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Neurocare Center for Research, Newton, Massachusetts
  - ClinSite, LLC, Ann Arbor, Michigan
  - Professional Clinical Research, Benzonia, Michigan
  - Hutzel Womens Health Research, Detroit, Michigan
  - Professional Clinical Research, Interlochen, Michigan
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Lawrence Ob-Gyn Assoc., PC, Lawrenceville, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - NY Center for Women's Health Research, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - Complete Healthcare for Women, Columbus, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - University Hospitals of Cleveland Landerbrook Health Center, Mayfield Heights, Ohio
  - Sooner Clinical Research, Inc., Oklahoma City, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Philadelphia Clinical Research, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Susan L Floyd, MD, PC, Wexford, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Tekton Research, Austin, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - Advances In Health, Inc., Houston, Texas
  - The Woman's Hospital of Texas Clinical Research Center, Houston, Texas
  - Research Across America, Katy, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Virginia Women's Center, Richmond, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
  - Tidewater Clinical Research, Inc, Virginia Beach, Virginia
  - Women's Clinical Research Center, Seattle, Washington
  - North Spokane Women's Clinic Research, Spokane, Washington

REFERENCES:
- [Derived] Pinkerton JV, Joffe H, Kazempour K, Mekonnen H, Bhaskar S, Lippman J. Low-dose paroxetine (7.5 mg) improves sleep in women with vasomotor symptoms associated with menopause. Menopause. 2015 Jan;22(1):50-8. doi: 10.1097/GME.0000000000000311. PMID 25137243
- [Derived] Portman DJ, Kaunitz AM, Kazempour K, Mekonnen H, Bhaskar S, Lippman J. Effects of low-dose paroxetine 7.5 mg on weight and sexual function during treatment of vasomotor symptoms associated with menopause. Menopause. 2014 Oct;21(10):1082-90. doi: 10.1097/GME.0000000000000210. PMID 24552977
- [Derived] Simon JA, Portman DJ, Kaunitz AM, Mekonnen H, Kazempour K, Bhaskar S, Lippman J. Low-dose paroxetine 7.5 mg for menopausal vasomotor symptoms: two randomized controlled trials. Menopause. 2013 Oct;20(10):1027-35. doi: 10.1097/GME.0b013e3182a66aa7. PMID 24045678
- See also: Sponsor — http://www.noven.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules: Subjects were randomized to receive Brisdelle (paroxetine mesylate) 7.5 mg Capsules administered orally once daily at bedtime beginning on Day 1 and continuing up to Day 84
- Placebo Capsules: Subjects were randomized to receive placebo capsules (sugar pill) orally administered once daily at bedtime beginning on Day 1 and continuing up to Day 84
Period: Overall Study
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Started | 306 | 308
Completed | 271 | 278
Not Completed | 35 | 30
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Physician Decision | 3 | 3
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 5 | 4
Not completed — Adverse Event | 8 | 4
Not completed — Eligibility Criteria Not Met | 2 | 3
Not completed — Failed C-SSRS | 5 | 2
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules; Placebo Capsules: Subjects were randomized to receive either Brisdelle (paroxetine mesylate) Capsules or placebo in a 1:1 ratio, administered once daily at bedtime beginning on Day 1 and continuing up to Day 84
- Total: Total of all reporting groups
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules | Total
Number analyzed (Participants) | 306 | 308 | 614
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 281 | 284 | 565
  >=65 years | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (5.95) | 54.5 (6.27) | 54.7 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306 | 308 | 614
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 306 | 308 | 614

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Frequency of Moderate to Severe VMS From Baseline at Week 4 and Week 12.
Description: Subjects recorded the number of hot flashes per week using an electronic diary. The results reported are not hot flashes per week.
  The results reported are:
  * Mean Baseline frequency of moderate to severe VMS
  * Mean change in frequency of moderate to severe VMS from baseline to Week 4
  * Mean change in frequency of moderate to severe VMS from baseline to Week 12.
Time Frame: Week 4 and Week 12
Population: The outcome data presented for these measurements were obtained using a scale questionnaire. Data were analyzed only from participants who completed and turned in the completed questionnaire. Therefore, the number of participants analyzed is not consistent with numbers provided in any of the rows in the participant flow module.
Measure: Mean (Standard Deviation); unit: Hot flash per day
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 301 | 305
Hot flash per day
  Baseline | 11.79 (4.87) | 11.65 (4.39)
  Week 4 | -4.71 (4.00) | -3.36 (4.65)
  Week 12 | -6.22 (4.53) | -5.33 (5.31)
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules vs Placebo Capsules; Test type: Superiority or Other; p < 0.0001, Rank transformed ANCOVA — Week 4 frequency
Statistical Analysis 2: Comparison: Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.0090, Rank transformed ANCOVA — Week 12 frequency

2. Secondary Outcome: Clinical Meaningfulness Anchored to Patient Global Improvement (PGI-I) (%)
Description: A patient improvement scale questionnaire was used during participant visits.
  The clinical meaningfulness of the observed treatment effect was demonstrated by performing the following analysis:
  Subjects were categorized in to 2 groups (satisfied and unsatisfied). Based on a 7 point patient global impression (PGI) questionnaire which assesses the subject improvement in VMS. Subjects were considered satisfied with their treatment if their response to the question "Compared to before starting the study medication, how would you describe your hot flushes now?" is 'Very much better' (1) or 'Much better' (2) or 'A little better' (3) and will be considered unsatisfied if their response to the same question is 'No change' (4) or 'A little worse' (5) or 'Much worse' (6) or 'Very much worse' (7). Receiver Operator Curve (ROC) analysis was performed on the combined data.
  Subjects who were satisfied with their treatment were considered to have a treatment effect with clinical meaningfulness
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of satisfied participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 301 | 305
Percentage of satisfied participants
  Week 4 | 50 | 37
  Week 12 | 51 | 43
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.001, Logit model — Clinical meaningfulness at week 4
Statistical Analysis 2: Comparison: Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.055, Logit model — Clinical meaningfulness at week 12

3. Secondary Outcome: Change From Baseline in Total Number of Awakenings Due to Hot Flashes, Median
Description: Participants completed a electronic diary to report nightime awakenings. Subjects took study drug once daily at bedtime and they were instructed to complete daily hot flash and sleep diaries to record the number of hot flashes daily, the severity of each episode of hot flash and total number of awakenings due to hot flashes.
  The diary data was used to evaluate and compare the treatment groups, on the change from baseline to Week 4 and Week 12, in the total number of awakenings due to hot flashes. The total number of awakenings due to hot flashes in the run-in period was used as baseline.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Nightime awakenings
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 289 | 288
Nightime awakenings
  Week 4 | -8.33 [-66.8 to 60.31] | -7.12 [-197.0 to 415.3]
  Week 12 | -12.00 [-66.8 to 63.31] | -11.05 [-197.0 to 29.83]

4. Secondary Outcome: Change in Frequency of Moderate to Severe Hot Flashes Frequency From Baseline (BMI <32 kg/m2, Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI <32 kg/m2 subgroup, the mean weekly reduction in frequency of moderate to severe hot flashes from Baseline was calculated for Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Hot flashes per week
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 211 | 206
Hot flashes per week
  Week 4 | -31.00 [-155 to 33.00] | -23.50 [-185 to 58.00]
  Week 12 | -46.00 [-163 to 84.00] | -35.00 [-189 to 50.00]

5. Secondary Outcome: Change in Frequency of Moderate to Severe Hot Flashes Frequency From Baseline (BMI ≥32 kg/m2, Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI ≥32 kg/m2 subgroup, the mean weekly reduction in frequency of moderate to severe hot flashes from Baseline was calculated for Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Hot flashes per week
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 77 | 87
Hot flashes per week
  Week 4 | -28.00 [-83 to 20.00] | -19.00 [-99 to 80.00]
  Week 12 | -35.00 [-115 to 40.00] | -37.50 [-180 to 44.00]

6. Secondary Outcome: Change in Severity of Moderate to Severe Hot Flashes From Baseline (BMI <32 kg/m2, At Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI <32 kg/m2 subgroup, the mean weekly reduction in the severity of moderate to severe hot flashes from Baseline was calculated at Week 4 and Week 12.
  Subjects recorded the number of hot flashes per week using an electronic diary. Severity score for hot flashes for each subject was calculated as the sum of 2 times the number of moderate hot flashes, plus 3 times the number of severe hot flashes, divided by the total number of moderate and severe hot flashes.
  Weekly Severity Score = (2•Fm +3•FS)/(Fm + FS) Daily Severity Score = {(2•F) m +3•FS)/(Fm + FS)}/7 Where, Fm= Frequency of Moderate Hot Flashes Fs = Frequency of Severe Hot Flashes The calculated severity score is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Hot Flash Severity scores per week
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 206 | 203
Hot Flash Severity scores per week
  Week 4 | -0.055 [-1.0 to 0.89] | 0.00 [-1.0 to 0.54]
  Week 12 | -0.043 [-.97 to 0.89] | -0.010 [-1.0 to 0.53]

7. Secondary Outcome: Change in Severity of Moderate to Severe Hot Flashes From Baseline (BMI ≥32 kg/m2, Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI ≥32 kg/m2 subgroup, the mean weekly reduction in the severity of moderate to severe hot flashes from Baseline was calculated at Week 4 and Week 12.
  Subjects recorded the number of hot flashes per week using an electronic diary. Severity score for hot flashes for each subject was calculated as the sum of 2 times the number of moderate hot flashes, plus 3 times the number of severe hot flashes, divided by the total number of moderate and severe hot flashes.
  Weekly Severity Score = (2•Fm +3•FS)/(Fm + FS) Daily Severity Score = {(2•F) m +3•FS)/(Fm + FS)}/7 Where, Fm= Frequency of Moderate Hot Flashes Fs = Frequency of Severe Hot Flashes The calculated severity score is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Hot Flash Severity scores per week
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 74 | 86
Hot Flash Severity scores per week
  Week 4 | -0.023 [-0.57 to 0.65] | -0.014 [-.081 to 0.43]
  Week 12 | -0.079 [-1.0 to 0.53] | -0.030 [-0.85 to 0.39]

8. Secondary Outcome: Change From Baseline in Greene Climacteric Scale (GCS) at Week 4 and Week 12, Total Score, Median
Description: The Greene Climacteric Scale (GCS) was used for this measurement. The scale has 21 questions and measures symptoms in 4 areas; these are psychological (anxiety and depression), physical, vasomotor, and libido.
  The severity of the symptom was scored as: 0=none, 1=mild, 2=moderate, and 3=severe. Anxiety was determined by using the sum of scores 1 to 6, and depression was determined by using the sum of scores 7 to 11. Physical aspects were determined by using the sum of scores 12 to 18; vasomotor aspects were determined by using the sum of scores 19 to 20; and libido was determined by using the score for question 21.
  The total GCS score ranges from "0" to "63" which is the sum of all the scores for the 21-symptom assessment questions in this scale. Each subject's total GCS score at baseline and at Week 4 and Week 12 were used to calculate change from baseline in these symptoms. The change from baseline is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 280 | 282
units on a scale
  Week 4 | -3.00 [-36.00 to 26.00] | -2.00 [-39.00 to 18.00]
  Week 12 | -4.00 [-36.00 to 49.00] | -3.00 [-44.00 to 24.00]

9. Secondary Outcome: Percentage of Responders
Description: Participants reported the number of hot flashes using an electronic diary. Participants who hd a ≥50% reduction in hot flash frequency were defined as responders. The percent of responders is presented below.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 301 | 305
percentage of participants
  Week 4 | 40.20 | 29.18
  Week 12 | 49.83 | 44.92

10. Secondary Outcome: Percentage of Patient Global Improvement (PGI) Scale Responders (%)
Description: Percentage of PGI Responders: Subject's overall improvement in VMS from baseline assessed using the Patient Global Improvement (PGI) scale. Responders: Subjects Achieving a Score of "Very Much Better" Or "Much Better" Or "A Little Better".
  Non Responders: Subjects with a Score of "No Change" Or "A Little Worse" Or "Much Worse" Or "Very Much Worse".
  Patient Global Improvement (PGI) scale is described below:
  Compared to before starting study medication, how would you describe your hot flushes now? 0 = Not assessed
  1. = Very much better
  2. = Much better
  3. = A little better
  4. = No change
  5. = A little worse
  6. = Much worse
  7. = Very much worse
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 301 | 305
percentage of participants
  Week 4 | 68.21 | 61.75
  Week 12 | 72.82 | 64.60

11. Secondary Outcome: Percent Daytime and Nighttime Responders, Numerical Rating Scale (NRS)
Description: Subject's overall improvement in VMS from Baseline assessed using the Numerical Rating Scale (NRS) The NRS is measured on a scale of 0 to 10 on how bothered the subject was by her VMS (0=not bothered at all and 10=very much bothered).
  The measure being reported below is percentage of responders who had an improvement in NRSscore at Week 4 and Week 12 compared to baseline. A responder is defined as a subject who had an improvement in the NRS score. An improvement is defined as a score ≤5 on each question.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 300 | 302
percentage of participants
  Week 4 | 39.00 | 30.46
  Week 12 | 46.51 | 45.72

12. Secondary Outcome: Change From Baseline in Arizona Sexual Experience Scale (ASEX, Week 4 and Week 12) Total Score
Description: The Arizona Sexual Experiences Scale (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction.
  The sum of the scores for all 5 items was calculated at Week 4 and Week 12. The results presented below are change from baseline at Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 280 | 282
units on a scale
  Week 4 | -0.34 (3.28) | -0.43 (2.87)
  Week 12 | -0.36 (3.77) | -0.61 (3.30)

13. Secondary Outcome: Effect of Paroxetine Mesylate Capsules on Percent Improvement of Hot Flash Interference From Baseline at Week 4 and Week 12, Hot Flash Related Daily Interference Scale (HFRDIS)
Description: Interference of hot flashes was measured by using the hot flash-related daily interference scale (HFRDIS). The HFRDIS is a 10-item scale that measures the degree to which hot flashes interfere with 9 daily activities and the tenth item measures the degree to which hot flashes interfere with each of the other items. Subjects can score for each item on a scale from 0 to 10 where 0 = Do not interfere and a score of 10 = Completely interferes.
  The measure being reported below is percentage of responders who had an improvement in HFRDIS score at Week 4 and Week 12 compared to baseline. A responder is defined as a subject who had an improvement in the HFRDIS score. An improvement is defined as a score ≤3 on each question.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 278 | 275
Percent of participants
  Week 4 | 26.98 | 32.00
  Week 12 | 19.67 | 21.95

14. Secondary Outcome: Percent Responders Improvement in VMS From Baseline Using the Clinical Global Impression (CGI) Scale.
Description: Proportion of NRS Responders: Subject's overall improvement in VMS from Baseline was assessed using the Numerical Rating Scale (NRS)
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  Responders: Subjects Achieving a Score of "Very Much Improved" Or "Much Improved" Or "Minimally Improved".
  Non Responders: Subjects with a Score of "No Change" Or "Minimally Worse" Or "Much Worse" Or "Very Much Worse".
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 280 | 285
percentage of participants
  Week 4 | 68.93 | 57.89
  Week 12 | 71.88 | 63.92

15. Secondary Outcome: Effect of Brisdelle (Paroxetine Mesylate) Capsules on Anxiety and Depression
Description: Depression & anxiety were measured by using the Hospital Anxiety & Depression Scale (HADS).
  The HADS was developed to assess anxiety & depression. It is meant to differentiate symptoms of depression with those of anxiety.
  Number of items: 14 (7 questions relating to anxiety; 7 questions relating to depression).
  Responses are based on the relative frequency of symptoms over the past week, using a four point scale ranging from 0 (not at all) to 3 (very often indeed).
  Responses are summed to provide separate scores for anxiety and depression symptomology with possible scores ranging from 0 to 21 for each scale.
  The results presented below are the percentage of participants with abnormal HADS Scores for both Abnormal Anxiety & Abnormal Depression at Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 281 | 281
Percentage of participants
  Week 4 | 3.56 | 3.56
  Week 12 | 2.02 | 2.75

16. Secondary Outcome: Assessment of Mood
Description: Mood was measured by using the Profile of Mood States (POMS) questionnaire. The Profile of Moods States (POMS) is a 65-item multi-dimensional measure that provides a method of assessing transient, fluctuating active mood states. Key areas that are measured include: tension-anxiety, anger-hostility, fatigue-inertia, depression-dejection, vigor-activity, confusion-bewilderment. Responses to questions are scored with the following numerical values: Not at all = 1, A little = 2, Moderate = 3, Quite a bit = 4, Extremely = 5. A total score for a domain was obtained by summing the responses of individual items in the domain. The total POMS score can range from "65" to "325." Each subject's total POMS score at baseline and at Week 4 and Week 12 were used to calculate the percent of participants with less disturbance in mood at Week 4 and Week 12 compared to baseline. The percent of participants with less disturbance in mood is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 280 | 280
Percent of participants
  Week 4 | 39.29 | 35.36
  Week 12 | 43.90 | 34.25

17. Secondary Outcome: BMI Change From Baseline (kg/m2), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  Assessment of the effect of Brisdelle compared with placebo on body mass index.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Change from baseline BMI kg/m2
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 282 | 288
Change from baseline BMI kg/m2
  Week 4 | 0.00 [-1.49 to 1.83] | 0.04 [-1.70 to 1.63]
  Week 12 | 0.00 [-2.16 to 2.58] | 0.17 [-7.44 to 2.58]

18. Primary Outcome: Mean Change From Baseline in Hot Flash Severity at Week 4 and Week 12
Description: Subjects recorded the number of hot flashes per week using an electronic diary. Severity score for hot flashes for each subject was calculated as the sum of 2 times the number of moderate hot flashes, plus 3 times the number of severe hot flashes, divided by the total number of moderate and severe hot flashes.
  Weekly Severity Score = (2•Fm +3•FS)/(Fm + FS) Daily Severity Score = {(2•F) m +3•FS)/(Fm + FS)}/7 Where, Fm= Frequency of Moderate Hot Flashes Fs = Frequency of Severe Hot Flashes The calculated severity score is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hot Flash Severity score per day
Arm/Group | Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules | Placebo Capsules
Number analyzed (Participants) | 301 | 305
Hot Flash Severity score per day
  Baseline | 2.528 (0.30) | 2.526 (0.31)
  Week 4 | -0.091 (0.25) | -0.046 (0.23)
  Week 12 | -0.104 (0.29) | -0.084 (0.29)
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.0017, Rank transformed ANCOVA — Week 4 severity
Statistical Analysis 2: Comparison: Brisdelle (Paroxetine Mesylate) 7.5 mg Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.1658, Rank transformed ANCOVA — Week 12 severity

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Serious Adverse Events (participants affected / at risk) | 2/301 | 1/305
Other Adverse Events (participants affected / at risk) | 134/301 | 129/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brisdelle (Paroxetine Mesylate) Capsules (N=301) | Placebo Capsules (N=305)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brisdelle (Paroxetine Mesylate) Capsules (N=301) | Placebo Capsules (N=305)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9) | 5 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Bloody discharge (General disorders) | 0 (0) | 1 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Energy increased (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (8) | 2 (2)
Influenza like illness (General disorders) | 1 (2) | 0 (0)
Irritability (General disorders) | 2 (2) | 4 (4)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Thirst (General disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Ear lobe infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (10) | 9 (9)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 11 (11)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 8 (8)
Urinary tract infection (Infections and infestations) | 6 (6) | 5 (5)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 2 (2)
Carotid bruit (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 2 (2) | 0 (0)
Haematocrit increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Food craving (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Crying (Nervous system disorders) | 0 (0) | 1 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (13) | 14 (17)
Hypersomnia (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 3 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 3 (3) | 0 (0)
Sedation (Nervous system disorders) | 2 (2) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Anorgasmia (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (4) | 3 (3)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Elevated mood (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (4)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 2 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 2 (2) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sweat gland disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Mole excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Scar excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other